CLINICAL TRIAL: NCT05602610
Title: Comprehensive Clinical and Laboratory Assessment of Visceral Leishmaniasis to Develop Clinical Prognostic Tools to Predict Relapse: a Prospective Cohort Study in Ethiopia
Brief Title: Clinical Prognostic Score to Predict Relapse in VL
Acronym: CPS
Status: Recruiting | Type: Observational
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: University of Gondar (Other)
Responsible Party: Sponsor
Other Study IDs: 1544/21
Record Dates: First submitted 2022-10-27; First posted 2022-11-02 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Visceral Leishmaniasis
Keywords: leishmaniasis; visceral; neglected; relapse; Ethiopia
MeSH Terms: conditions — Leishmaniasis, Visceral; Leishmaniasis; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, tissue, sputum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- VL patients: VL infected individuals residing in/ with travel history to VL-endemic areas in Northern Ethiopia
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This prospective cohort study has the aim to develop a prognostic tool to predict relapse in patients suffering from visceral leishmaniasis (VL) from VL endemic regions in Ethiopia.

Therefore, comprehensive clinical and laboratory characterization of all confirmed VL patients before and during treatment will be performed in order to identify the factors that determine prognosis of the patients. This approach would result in more efficient patient care and would reduce the case fatality and morbidity, and improve follow-up and care for those at risk of VL relapse.

DETAILED DESCRIPTION:
Certain patient groups seem to be at higher risk of poor outcomes. Although the average case fatality rate was <10% in Ethiopia , certain subgroups of VL patients are at significantly higher risk of dying, with case fatality rates as high as 39% when patients coinfected with HIV or sepsis. The host's immunocompetence appears to play a critical factor associated with disease development, severity, treatment success and disease relapse. Yet, a substantial group of immunocompetent patients also fail to respond well to treatment, or develop relapse after cure. Relapse is increasingly recognized as an important clinical challenge, with 10-15% estimated to develop relapse in the Ethiopian setting. Understanding which factors determine prognosis among VL patients is key in improving outcomes, as high-risk patients can be identified and receive additional monitoring, care, investigations or preferential treatment with safer or more effective drugs.

One of the strategies to improve patient outcome is identification of factors that determine the prognosis of a patient. These factors can be used in clinical decision tools to provide the most appropriate care for each patient. With the key prognostic factors, patients can be stratified in high and low risk of relapse, treatment failure and mortality and can be treated accordingly, providing intensive monitoring and/or treatment of comorbidities of high-risk patients and a more decentralized follow-up for low-risk patients. This approach would result in more efficient patient care and would reduce the case fatality and morbidity, and improve follow-up and care for those at risk of VL relapse.

No clinical tools for prediction of relapse and treatment failure currently exist. The existing clinical tools for predicting mortality developed so far have a fair accuracy but these tools could further be improved by using prognostic markers both before and during treatment and including more relevant parameters which were previously ignored, such as more laboratory parameters including coagulation profile, blood culture, immunological markers and more relevant clinical parameters such as sepsis and comorbidities.

This study will perform a comprehensive clinical and laboratory characterization of all confirmed VL patients before and during treatment with the main objective to develop a prognostic tool for unfavorable outcome among hospitalized patients. It is planned to develop tools of different complexity, geared towards the capacity of the health facility and also study the added effect of each variable in the tool. The data from this study will address a number of outstanding unanswered questions that could help to improve or standardize VL management.

ELIGIBILITY:
Inclusion Criteria:

* clinically or parasitologically confirmed VL

Exclusion Criteria:

* Age under 12 years
* VL patients already on treatment for 3 days or more
* Severe critical condition or other circumstances that make the study medically inadvisable
* Unlikely to adhere to follow up visits during the study period (e.g. patients who live or work very far away) AND not reachable by phone for follow-up information
* Pregnant or lactating woman

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with clinically or parasitologically confirmed VL in Northern Ethiopia
Sampling Method: Probability Sample
Enrollment: 741 (Estimated)
Dates: Start 2023-02-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Identification of risk factors for relapse | December 2026
  The association between development of relapse and potential risk factors (demographic/clinical characteristics as well as host immunity/Leishmania infection markers)
Prognostic tool for relapse | December 2026
  A clinical decision algorithm, prioritizing and integrating identified risk factors, that is able to most efficiently predict the risk of developing relapse within 12 months after start of treatment

SECONDARY OUTCOMES:
Patterns in host immune markers for VL relapse, treatment failure and death | December 2026
  The association between the risk of VL relapse/ treatment failure/ death and the levels and evolution of the different host immune markers.
Identification of risk factors for treatment failure | December 2026
  The association between the occurence of treatment failure and potential risk factors (demographic/clinical characteristics as well as host immunity/Leishmania infection markers)
Identification of risk factors for death | December 2026
  The association between occurrence of death and potential risk factors (demographic/clinical characteristics as well as host immunity/Leishmania infection markers)

CONTACTS AND LOCATIONS:
Overall Officials: Saskia van Henten, MD, Study Chair — Institute of Tropical Medicine Antwerp, Antwerp, Belgium; Eleni Ayele, MD, Principal Investigator — University of Gondar, Gondar, Ethiopia
Locations (1):
- University of Gondar, Gonder, Ethiopia

IPD SHARING:
Plan to Share IPD: Undecided
Raw data may be made available through a controlled access procedures (privacy restrictions)